CLINICAL TRIAL: NCT04069026
Title: An Open-label, Phase 1, First-in-human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics and Tumor Response Profile of the Aryl Hydrocarbon Receptor Inhibitor (AhRi) BAY 2416964 in Participants With Advanced Solid Tumors
Brief Title: A First-in-Humans Dose Finding Study for an Aryl Hydrocarbon Receptor Inhibitor (AhRi) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20201; 2023-503546-32-00 (Other: CTIS (EU)); 2019-000722-22 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-08-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumors
Keywords: Non-small cell lung cancer (NSCLC); Head and neck squamous cell carcinoma (HNSCC); Advanced cancer; Immunotherapy; Immuno oncology; Aryl Hydrocarbon Receptor inhibitor(AhRi); Aryl Hydrocarbon Receptor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation of BAY2416964 (Experimental): Approximately 8 dose levels of BAY2416964 are planned
  Interventions: Drug: BAY2416964
- Dose expansion of BAY2416964 in tumor type specific (Experimental): Patients with NSCLC, HNSCC
  Interventions: Drug: BAY2416964

INTERVENTIONS:
Drug: BAY2416964 — Oral application of study drug daily in a predefined dose escalation scheme.
  Arms: Dose escalation of BAY2416964
Drug: BAY2416964 — Oral application of study drug daily at the dose defined in the dose escalation scheme to determine the recommended phase 2 dose (RP2D).
  Arms: Dose expansion of BAY2416964 in tumor type specific

SUMMARY:
In this study researchers want to gather relevant information regarding the safety of BAY2416964 and how well the drug works in participants with a type of solid tumors that cannot be cured by currently available drugs. Researchers want to find the highest dose of BAY2416964 that participants could take without having too many side effects, how the drug is tolerated and the way the body absorbs, distributes and gets rid of the study dug. BAY2416964 is a small molecule which blocks the Aryl Hydrocarbon Receptor (a protein involved in immune cell reaction to tumor cells) allowing the body to use its immune response against the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age inclusive, at the time of signing the informed consent.
* Participants with following histologically or cytologically confirmed advanced solid tumors that have progressed after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment.

  * Dose Escalation: all solid tumor types
  * Tumor type-specific high-dose (MTD or MAD) Expansion cohorts: Will be grouped by tumor type:

    * NSCLC
    * HNSCC
  * NSCLC (TID dosing) expansion cohorts
* Have measurable disease per RECIST 1.1 as assessed by CT/MRI. At least one measurable lesion by RECIST 1.1 is required. Lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered measurable if progression has been demonstrated in such lesions.
* Life expectancy at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG)performance status of 0 to 1.
* Adequate bone marrow and organ function as assessed by the following laboratory tests performed within 7 days before treatment initiation.

  * Bone marrow reserve:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    * Hemoglobin (Hb) ≥ 9.0g/dL, without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
    * Platelet count ≥ 100 x 10^9/L. Transfusion to meet the inclusion criteria will not be allowed.
  * Hepatic:

    * Total bilirubin ≤ 1.5 x the upper limit of normal range (ULN). Known Gilbert syndrome is allowed if total bilirubin is ≤ 3 x ULN.
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases).
    * Albumin > 25 g/L.
  * Renal:

    --- eGFR ≥ 60 mL/min as calculated using the MDRD equation or creatinine level ≤ 1.5x ULN.
  * Lipase and amylase ≤ 1.5 x ULN.
  * Coagulation:

    * International normalized ratio (INR) OR prothrombin time (PT) AND activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless the participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* Adequate cardiac function, measured by echocardiography within 28 days before start of study intervention (left ventricular ejection fraction within institutional normal range for age and gender).

Exclusion Criteria:

* Severe (CTCAE v.5 Grade ≥ 3) infections within 4 weeks before the first BAY2416964 administration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia. Clinically active infections (CTCAE v.5 > Grade 1) within 2 weeks before the first BAY2416964 administration.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) within 1 week before the first dose of study intervention or any other form of immunosuppressive therapy within 2 weeks prior the first dose of study intervention.
* Congestive heart failure New York Heart Association (NYHA) greater than Class I or cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or calcium channel blockers.
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis.

Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that repeat imaging needs to be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.

* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Significant acute gastrointestinal disorders with diarrhea as a major symptom, e.g. Crohn's disease, malabsorption, or ≥ NCI-CTCAE v. 5.0 Grade 2 diarrhea of any etiology.
* History of organ allograft transplantation, including allogeneic bone marrow transplantation.
* Has received prior radiotherapy within 2 weeks before start of BAY2416964 or received radiation therapy to the lung that is > 30 Gy within 6 months before start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Treatment with systemic immunosuppressant medications (including but not limited to

  * > 10 mg/day prednisone or equivalent within 1 week before the first study intervention administration.
  * any other form of immunotherapy, e.g., cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks before the first BAY2416964 administration.

The use of inhaled corticosteroids, or low doses of glucocorticoids (no more than 10 mg/day prednisone or equivalent; if a higher dose would be needed to maintain adrenal function investigator must obtain approval from sponsor), and mineralocorticoids (e.g. fludrocortisone for adrenal insufficiency) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment emergent adverse events (TEAEs) including treatment-emergent serious adverse events (TESAEs) and dose-limiting toxicities (DLTs) | Up to 90 days after end of treatment
Severity of treatment emergent adverse events (TEAEs) including treatment-emergent serious adverse events (TESAEs) and dose-limiting toxicities (DLTs) | Up to 90 days after end of treatment
Maximum tolerated dose (MTD) or maximum administered dose (MAD) of BAY2416964 | Cycle 1 (21 days) in dose escalation
  MTD:defined as the dose level that can be given such that the estimated Dose limiting toxicity (DLT) probability is closest to approximately 25%.
Recommended Phase II dose (RP2D) of BAY2416964 | Up to 90 days after end of treatment
  Integration of all available safety, PK and PD data
Maximal plasma exposure (Cmax) for once daily (QD) dosing of BAY2416964 after single-dose and multiple-dose in Cycle 1. | From pre-dose up to 24 hours after administration on Cycle 1 (21 days) Day 1. From pre-dose up to 12 hours after administration on Cycle 1 (21 days) Day 15
Area under the curve [AUC (0 - t)] (t=6,12 or 24 dependent on the dosing regimen) of BAY2416964 after single and multiple-dose in Cycle 1 | From pre-dose up to 6, 12, or 24 hours after administration on Day 1 and/or Day 15 in Cycle 1 (21 days).

SECONDARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | At the end of Cycle 2 (- 7 days), Cycle 4 (-7 days), every 9 weeks (- 7 days) from Cycle 5 to Cycle 10 and every 4th cycle (- 7 days) from Cycle 11 onwards. Each cycle is 21 days.
Change from baseline in AhR target gene expression in whole blood after ex-vivo stimulation | Screening, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 4 Day 1(each cycle is 21 days)
Cytokine measurements, e.g. IL-6 (immunoassay), in whole blood after ex-vivo stimulation. | Screening, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 4 Day 1(each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - Yale University School of Medicine, New Haven, Connecticut
  - Greenville Health System, Greenville, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics | START San Antonio, San Antonio, Texas
- Canada (2):
  - Princess Margaret Hospital-University Health Network, Toronto, Ontario
  - CHU de Québec-Hôpital de l'Enfant-Jésus, Québec
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Charité Campus Benjamin Franklin (CBF), Berlin
- Spain (5):
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Ramón y Cajal | Oncología, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria | Cardiology Department, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.